CLINICAL TRIAL: NCT00144989
Title: A Phase III Study Comparing Etoposide and Cisplatin (EP) With Irinotecan and Cisplatin (IP) Following EP Plus Concurrent Accelerated Hyperfractionated Thoracic Irradiation (EP/TRT) for Limited-Stage Small-Cell Lung Cancer : JCOG0202-MF
Brief Title: A Study Comparing Irinotecan and Cisplatin (IP) With Etoposide and Cisplatin (EP) Following EP/TRT for LD-SCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0202-MF; C000000095
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Small-Cell-Lung Cancer
Keywords: Small-cell lung cancer; Limited-Stage Small-Cell Lung Cancer; Combined modality therapy; chemotherapy; radiotherapy; Irinotecan; Cisplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Etoposide and cisplatin after chemoradiotherapy
  Interventions: Drug: Etoposide and cisplatin after chemoradiotherapy
- 2 (Experimental): Irinotecan and cisplatin after chemoradiotherapy
  Interventions: Drug: Irinotecan and cisplatin after chemoradiotherapy

INTERVENTIONS:
Drug: Etoposide and cisplatin after chemoradiotherapy — Etoposide and cisplatin after chemoradiotherapy
  Arms: 1
Drug: Irinotecan and cisplatin after chemoradiotherapy — Irinotecan and cisplatin after chemoradiotherapy
  Arms: 2

SUMMARY:
To evaluate the role of 3 cycles of irinotecan and cisplatin for patients with limited-stage small-cell lung cancer who received one course of etoposide and cisplatin plus concurrent accelerated hyperfractionated thoracic irradiation.

DETAILED DESCRIPTION:
The Japan Clinical Oncology Group (JCOG) previously conducted a randomized phase III trial comparing irinotecan and cisplatin (IP) with EP in patients with extensive-stage SCLC. The response rate and overall median survival were significantly better for IP, i.e. 84.4% and 12.8 months with IP, versus 67.5% and 9.4 months with EP, respectively. The 2-year survival rates were 19.5% for IP and 5.2% for EP (7). These encouraging results prompted us to explore the use of IP in LSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. cytologically, histologically proven small-cell lung cancer
2. limited disease
3. age 20-70 years old
4. performance status of 0-1
5. measurable disease
6. no prior treatment for small-cell lung cancer
7. no history of chemotherapy
8. adequate organ functions
9. written informed consent

Exclusion Criteria:

1. pericardial effusion
2. active concomitant malignancy
3. pregnant or lactating women
4. interstitial pneumonia/active lung fibrosis on chest x-ray, watery diarrhea, intestinal obstruction or paralysis, uncontrolled heart disease or a history of myocardial infarction within the previous 6 months, uncontrolled diabetes mellitus, active infection, psychological disease deemed unacceptable for inclusion to the study, long-term steroid treatment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2002-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
overall survival | during the study conduct

SECONDARY OUTCOMES:
adverse events of induction chemoradiotherapy | during the study conduct
chemotherapy after chemoradiotherapy | during the study conduct
late radiation morbidity | during the study conduct
serious adverse event | during the study conduct
progression-free survival | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Nishiwaki, MD, Study Chair — National Cancer Center Hospital East
Locations (37):
- Japan (37):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, Okazaki,Kake-machi,Kuriyado,18, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kyushu University Hospital, Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Gifu Municipal Hospital, Gifu,Kashima-cho,7-1, Gifu
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - National Nishigunma Hospital, Shibukawa,Kanai,2854, Gunma
  - National Hospital Organization, Dohoku National Hospital, Asahikawa,Hanasaki,7-4048, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo,Shiroishi-ku,Kikusui,4-2-3-54, Hokkaido
  - Hyogo Medical Center for Adults, Akashi,Kitaouji-cho,13-70, Hyōgo
  - Kobe City General Hospital, Kobe,Chuo-ku,Minatojimanakamachi,4-6, Hyōgo
  - Hyogo College of Medicine, Nishinomiya,Mukogawa-cho,1-1, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Yokohama Mucipical Citizen's Hospital, Yokohama,Hodogaya-ku,Okazawa-cho,56, Kanagawa
  - Kumamoto Regional Medical Center Hospital, Kumamoto,Honjo,5-16-10, Kumamoto
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Okayama University Hospital, Okayama,Shikata-cho,2-5-1, Okayama-ken
  - Osaka Prefectural Medical Center for Respiratory and Allergic Disease, Habikino,Habikino,3-7-1, Osaka
  - Rinku General Medical Center, Izumisano,rinku-ohrai-kita,2-23, Osaka
  - Graduate School of Medicine, Osaka City University, Osaka,Abeno-ku,Asahi-machi,1-5-7, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Osaka General Medical Center, Osaka,Sumiyoshi-ku,Bandai-higashi,3-1-56, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai,Nagasone,1180, Osaka
  - National Hospital Organization Toneyama National Hospital, Toyonaka,Toneyama,5-1-1, Osaka
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - Toranomon Hospital, Minato-ku,Toranomon,2-2-2, Tokyo
  - International Medical Center of Japan, Shinjuku-ku,Toyama,1-21-1, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- [Derived] Kubota K, Hida T, Ishikura S, Mizusawa J, Nishio M, Kawahara M, Yokoyama A, Imamura F, Takeda K, Negoro S, Harada M, Okamoto H, Yamamoto N, Shinkai T, Sakai H, Matsui K, Nakagawa K, Shibata T, Saijo N, Tamura T; Japan Clinical Oncology Group. Etoposide and cisplatin versus irinotecan and cisplatin in patients with limited-stage small-cell lung cancer treated with etoposide and cisplatin plus concurrent accelerated hyperfractionated thoracic radiotherapy (JCOG0202): a randomised phase 3 study. Lancet Oncol. 2014 Jan;15(1):106-13. doi: 10.1016/S1470-2045(13)70511-4. Epub 2013 Dec 3. PMID 24309370
- See also: Related Info — http://www.jcog.jp/